CLINICAL TRIAL: NCT05063604
Title: Randomized, Controlled, Open and Unicentric Phase II Clinical Trial, With Two Parallel Groups, to Evaluate the Antidepressant Efficacy of Psychotherapy and Citalopram in Women Diagnosed With Breast Cancer and Major Depression
Brief Title: Antidepressant Efficacy of Psychotherapy and Citalopram in Patients With Breast Cancer and Major Depression
Acronym: CAMAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The CAMAD clinical trial has been terminated due to difficulties in recruiting patients.
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Cinto Segalàs Cosi, MD, Psychiatrist at the Bellvitge University Hospital. Researcher at the Bellvitge Biomedical Research Institute (IDIBELL). Associate professor at the Clinical Sciences Department of the Barcelona University (UB)., Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-PSI-CAMAD; 2019-004548-31 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-10-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Major Depressive Episode
Keywords: Breast Cancer; Major Depressive Episode; Antidepressant Efficacy; Psychotherapy; Citalopram
MeSH Terms: conditions — Breast Neoplasms | interventions — Citalopram; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citalopram 20-40 mg (Experimental): Participants received citalopram 20 mg tablet once or twice daily for 12 weeks.
  Interventions: Drug: Citalopram
- Psychotherapy (Experimental): Participants received one psychotherapy session weekly for 12 weeks.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Citalopram — 20 mg tablet one or twice daily for 12 weeks
  Other Names: Prisdal
  Arms: Citalopram 20-40 mg
Behavioral: Psychotherapy — One session weekly for 12 weeks
  Arms: Psychotherapy

SUMMARY:
To provide evidence on the antidepressant efficacy of two therapeutic treatments: pharmacological treatment (citalopram) and psychotherapy treatment, in women diagnosed with breast cancer and major depression.

ELIGIBILITY:
Inclusion Criteria:

* Female patients first time diagnosed with breast cancer (stage I, II, III, or IV) between ages 18 and 75 (both inclusive).
* Patients with a "moderate-severe" level of emotional distress who meet the diagnostic criteria for major depression for at least two weeks or adjustment disorder with depressive mood for at least two months, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria (DSM-V), during the twelve months following the diagnose of breast cancer.
* Informed Consent Form Signature

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Suicide risk.
* Metastatic brain disease.
* Personal History of oncological disease.
* Personal History of serious somatic disease (cardiac, hepatic, respiratory, endocrinological, neurological and haematological).
* Personal History of organic brain disorder, substance abuse/dependence.
* Personal History of psychotic disorder, bipolar disorder and/or mental retardation.
* Contraindications of citalopram treatment.
* Taking antidepressants after the breast cancer diagnosis.
* Psychotherapy treatment after breast cancer diagnosis .

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in severity of depression on the Beck Depression Inventory (BDI) at week 12. | Every three weeks from baseline to the end of the study at week 12 (5 assessments in total).
  The BDI is a validated, self-reported instrument assessing the severity of depression. Scoring range 0-9 indicates minimal depression, 10-18 mild depression, 19-29 moderate depression, and 30-63 severe depression.

SECONDARY OUTCOMES:
Change from Baseline in quality of life on the European Quality of Life Scale Five Dimensions and Three Levels (EQ-5D-3L) at week 12. | Baseline and week 12.
  The EQ-5D-3L is a standardized measure of health-related quality of life. The EQ-5D descriptive system comprises five dimensions with three levels of severity: 1 indicates no problems, 2 some problems, and 3 extreme problems.
Change from Baseline in social-labor adaptation measured by number of days off work at week 12. | Every three weeks from baseline to the end of the study at week 12 (5 assessments in total).
  Number of days off work.
Age of patients. | Baseline.
  Measured in years.
Marital status. | Baseline.
  Percentage of patients single, married, widowed, separated or divorced collected by a clinical interview.
Cancer treatment received. | Baseline.
  Percentage of patients treated with surgery, radiotherapy, chemotherapy and/or hormonal therapy. This treatment information will be collected from the medical record.
Breast cancer stage. | Baseline.
  Breast cancer stage is expressed as a number on a scale from 0 to IV, where 0 describes non-invasive cancers that remain within their original location, and IV describes invasive cancers that have spread outside the breast to other parts of the body. This clinical information will be collected from the medical record.
Basal whole-brain activity by performing a functional Magnetic Resonance Imaging (fMRI). | fMRI at baseline.
  fMRI is a specialized form of magnetic resonance imaging used to examine regional brain activity, allowing the identification of the brain areas allegedly underpinning psychological processes. fMRI uses a specific imaging sequence (echo planar imaging) to measure small changes in blood oxygenation by assessing the so-called blood oxygenation level dependent (BOLD) signal over time, which is linked to regional neuronal function.
Change from baseline in emotional processing on the Dot-Probe Task (DPT). | DPT at baseline and week 12.
  The DPT is a validated task to assess emotional processing by measuring reaction time to two types of stimuli (emotional face vs. neutral face), each one displayed on a different side of the screen. A faster reaction to emotional stimuli than to neutral ones indicates a bias of attention towards the emotional face and reflects dysfunction on emotional processing.
Cost-effectiveness ratio differences between pharmacological treatment with citalopram and psychological treatment in patients in our environment with breast cancer (BC) and major depression (MD). | At week 12.
  Analyze the cost of several variables, including both treatments (pharmacological and psychological), use of infrastructures and travel costs (only the first inclusion visit will be in person, the subsequent follow-up will be online).
Number and severity of secondary side effects related to the consumption of pharmacological treatment with citalopram according to the side effects rating scale Udvalg für Kliniske Undersogelser (UKU). | At week 3, 6, 9 and 12.
  The UKU side effects scale is designed to evaluate the secondary effects derived from the consumption of psychotropic drugs. The UKU scale comprises a total of 54 items that describe 54 side effects. Each item takes a value from 0 to 3 (0, no or doubtful present; 1, mild; 2, moderate; 3, severe).

CONTACTS AND LOCATIONS:
Overall Officials: Cinto Segalàs, MD, PhD., Principal Investigator — Psychiatrist at the Bellvitge University Hospital.
Locations (1):
- Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fann JR, Thomas-Rich AM, Katon WJ, Cowley D, Pepping M, McGregor BA, Gralow J. Major depression after breast cancer: a review of epidemiology and treatment. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):112-26. doi: 10.1016/j.genhosppsych.2007.10.008. PMID 18291293
- [Result] Vodermaier A, Linden W, Rnic K, Young SN, Ng A, Ditsch N, Olson R. Prospective associations of depression with survival: a population-based cohort study in patients with newly diagnosed breast cancer. Breast Cancer Res Treat. 2014 Jan;143(2):373-84. doi: 10.1007/s10549-013-2795-4. Epub 2013 Dec 13. PMID 24337537
- [Result] Miguel C, Albuquerque E. Drug interaction in psycho-oncology: antidepressants and antineoplastics. Pharmacology. 2011;88(5-6):333-9. doi: 10.1159/000334738. Epub 2011 Nov 26. PMID 22123153
- [Result] Ochoa, C., & Casellas-Grau, A. (2015). Positive Psychotherapy in Cancer: Facilitating Posttraumatic Growth in Assimilation and Accomodation of Traumatic Experience. In C.R. Martin, V. R. Preedy & B. P.Vinood (Eds.). Comprehensive Guide to Post-Traumatic Stress Disorder (pp.113-127). Verna: Springer International Publishing Switzerland.
- [Result] Godlewska BR, Browning M, Norbury R, Igoumenou A, Cowen PJ, Harmer CJ. Predicting Treatment Response in Depression: The Role of Anterior Cingulate Cortex. Int J Neuropsychopharmacol. 2018 Nov 1;21(11):988-996. doi: 10.1093/ijnp/pyy069. PMID 30124867
- [Result] Victor TA, Furey ML, Fromm SJ, Ohman A, Drevets WC. Relationship between amygdala responses to masked faces and mood state and treatment in major depressive disorder. Arch Gen Psychiatry. 2010 Nov;67(11):1128-38. doi: 10.1001/archgenpsychiatry.2010.144. PMID 21041614
- [Result] Victor TA, Furey ML, Fromm SJ, Ohman A, Drevets WC. Changes in the neural correlates of implicit emotional face processing during antidepressant treatment in major depressive disorder. Int J Neuropsychopharmacol. 2013 Nov;16(10):2195-208. doi: 10.1017/S146114571300062X. Epub 2013 Jul 1. PMID 23809145
- [Result] Avis NE, Levine B, Naughton MJ, Case LD, Naftalis E, Van Zee KJ. Age-related longitudinal changes in depressive symptoms following breast cancer diagnosis and treatment. Breast Cancer Res Treat. 2013 May;139(1):199-206. doi: 10.1007/s10549-013-2513-2. Epub 2013 Apr 16. PMID 23588951
- [Result] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- See also: Citalopram technical data sheet. — http://cima.aemps.es/cima/pdfs/es/ft/60884/FT_60884.html.pd

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT05063604/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05063604/ICF_001.pdf